CLINICAL TRIAL: NCT05423509
Title: Dynamic Myofascial and Articular Mobilization and Reorganization (DMAMR) Treatment in Adolescent Idiopathic Scoliosis (AIS)
Brief Title: Myofascial and Articular Treatment of Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Selina Silva, Associate Professor, Orthopaedic Surgerey, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Study 20-228
Record Dates: First submitted 2022-06-01; First posted 2022-06-21 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Scoliosis Idiopathic Adolescent Treatment
Keywords: scoliosis; adolescent; chiropractor; myofascial; idiopathic
MeSH Terms: conditions — Scoliosis | interventions — Observation; Braces

STUDY DESIGN:
Intervention Model Description: randomized controlled trial between 2 treatment groups
Who Masked: Outcomes Assessor
Masking Description: The follow-up visits were performed by an advanced practice provider that did not know which treatment arm the patient is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment for AIS (Other): These are the participants with AIS that recieved the standard treatment with observation or bracing depending on the size of their curve.
  Interventions: Other: Standard AIS treatment with observation or bracing
- Treatment with Dynamic Myofascial Manipulation (Experimental): These are the participants that still received the standard treatment with observation or bracing depending on the size of their curve, but also had weekly treatment with a chiropractor for 6 months for dynamic myofascial manipulation
  Interventions: Other: Dynamic myofascial manipulation; Other: Standard AIS treatment with observation or bracing

INTERVENTIONS:
Other: Dynamic myofascial manipulation — Dynamic myofascial manipulation of the muscles in the back to improve the scoliosis appearance/flexibility/rotation
  Arms: Treatment with Dynamic Myofascial Manipulation
Other: Standard AIS treatment with observation or bracing — Observation with radiographs and bracing of curves greater than 20 degrees

SUMMARY:
Randomized controlled trial of participants with scoliosis into standard treatment with observation/bracing and the other group will have the added treatment of dynamic myofascial manipulation for 6 months.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a pilot study of the Dynamic Myofascial and Articular Mobilization and Reorganization (DMAMR) treatment in Adolescent Idiopathic Scoliosis (AIS). The investigators propose the implementation of Dynamic Myofascial and Articular Mobilization and Reorganization (DMAMR) protocol can (a) decrease and/or reduce progression of spinal curvatures, (b) reduce degree of anatomical rib hump deformity common in AIS, (c) decrease incidence of patients requiring corrective bracing and/or corrective spinal surgery, (d) significantly reduce AIS-associated pain, and (e) improve quality of life for AIS participants.

This study will test whether DMAMR produces clinically relevant changes in progression of scoliosis curvatures and rib humps, and whether this treatment protocol improves pain scores and quality of life.

Current research has demonstrated unilateral muscle shortening in AIS. Of most importance for this research proposal, research has also identified a set of muscles, portions of which are at an angle to the spine, that are shorter on the concave side of the curvature: the quadratus lumborum, psoas major and minor, and the abdominal obliques. The researchers have suggested this is a compensatory effect of the spinal deformities seen1. The investigators agree that unilateral muscle shortening is present in AIS but the investigators suggest that this asymmetry represents differences between muscle tension on either side of the spine and results in a tethering effect on the spine itself. Supporting a finding of the importance of these muscle imbalances, research using individualized physical therapeutic exercise programs to balance these types of muscle imbalances has demonstrated effectiveness in AIS treatment.

The investigators hypothesize this asymmetrical muscle imbalance, and its resultant tethering effect on the spine, represent myofascial dysfunction. The investigators believe the forces generated by this dysfunction are sufficient to induce worsening of the AIS curvature. The myofascial factors involved in the tethering of the spine in AIS include asymmetrical muscle imbalances involving muscles at an angle to the spine, primarily iliopsoas, quadratus lumborum, abdominal obliques, latissimus dorsi, and anterior serratus muscles.

Fascia overlies and interpenetrates these muscles. At a critical point, these myofascial imbalances generate sufficient stress on the overlying fascia to create a further contractile force within the fascia itself. The investigators ask whether this contractile force is mediated not only by anatomic shortening of individual muscle groups but also by intrinsic changes in fibroblast gene expression within the fascia itself.

The investigators further hypothesize that the asymmetrical muscle imbalances observed in AIS may be part of a larger contracted fascial spiral force influencing the development and progression of deformity. Therefore, treatment of the muscles, fascia, and related articular dysfunction may contribute to the control or reduction of AIS-associated deformities including scoliotic curvatures and accompanying rib humps. Effective treatment of these imbalances and deformities may reduce or eliminate AIS-associated spinal area pain, which the investigators hypothesize is largely myofascial in nature.

ELIGIBILITY:
Inclusion Criteria:

* Age from 10-15
* Scoliosis curve of 15-30 degrees on cobb angle
* Risser stage of 0-2

Exclusion Criteria:

* outside of age range, cobb angle or maturity level

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-06-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UNM Carrie Tingley Hospital, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment for AIS: These are the participants with AIS that received the standard treatment with observation or bracing depending on the size of their curve.
  Standard AIS treatment with observation or bracing: Observation with radiographs and bracing of curves greater than 20 degrees
Period: Overall Study
Arm/Group | Standard Treatment for AIS | Treatment With Dynamic Myofascial Manipulation
Started | 9 | 12
Completed | 9 | 10
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Standard Treatment for Adolescent Idiopathic Scoliosis: These are the participants with Adolescent Idiopathic Scoliosis that received the standard treatment with observation or bracing depending on the size of their curve.
  Standard AIS treatment with observation or bracing: Observation with radiographs and bracing of curves greater than 20 degrees
- Total: Total of all reporting groups
Arm/Group | Standard Treatment for Adolescent Idiopathic Scoliosis | Treatment With Dynamic Myofascial Manipulation | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 12 | 21
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 12.5 [10 to 15] | 12.5 [10 to 15] | 12.5 [10 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Cobb Angle
Description: Cobb angle as measured on x-ray
Time Frame: At time of enrollment
Population: We did not have as many patients enroll as originally expected because of COVID
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Standard Treatment for AIS | Treatment With Dynamic Myofascial Manipulation
Number analyzed (Participants) | 9 | 12
degrees | 18.9 [15 to 23] | 23.8 [14.6 to 33]

2. Primary Outcome: Cobb Angle
Description: Cobb angle as measured on x-ray
Time Frame: 6 months from time of enrollment
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Standard Treatment for AIS | Treatment With Dynamic Myofascial Manipulation
Number analyzed (Participants) | 9 | 12
degrees | 21.3 (6.3) | 25.3 (12.9)

3. Primary Outcome: Scoliometer Degree
Description: The degree of rotation measured clinically with a scoliometer
Time Frame: At time of enrollment
Population: We did not have the scoliosis reading on one patient in the beginning visit for the control group.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Standard Treatment for AIS | Treatment With Dynamic Myofascial Manipulation
Number analyzed (Participants) | 8 | 12
degrees | 7.4 (3.3) | 8.1 (4.4)

4. Primary Outcome: SRS-22
Description: The SRS-22 or Scoliosis Research Society-22 is a functional survey for the patient to fill out on their scoliosis. This survey has been validated in the literature. It is a 22 question survey on the functional status and pain that a patient experiences. Created by the scoliosis research society. There is a scoring rubric that goes with the survey. This survey has 5 domains that are covered with the minimum score of 22 and the maximum score of 110. The higher the score the better the patient is doing in the domains of: Activities of Daily Living, Mental Health, Pain, Patient Satisfaction, Positive Affect, Quality of Life, Social Relationships, and Stress/Coping.
Time Frame: At time of enrollment
Population: This is the number of participants in each group and the outcome measure numbers represent the baseline or SRS-22 scores at the time of enrollment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment for AIS | Treatment With Dynamic Myofascial Manipulation
Number analyzed (Participants) | 9 | 12
units on a scale | 84.2 (10.1) | 85.1 (11.8)

5. Primary Outcome: SRS-22
Description: as for outcome 4
Time Frame: 6 months from time of enrollment
Population: This is their SRS-22 scores 6 months into the study for each treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment for AIS | Treatment With Dynamic Myofascial Manipulation
Number analyzed (Participants) | 8 | 10
units on a scale | 80.9 (10.2) | 89.1 (8.6)

6. Primary Outcome: Pain Scale
Description: Question asking each participant about their back pain level using a visual analog scale of 0-10. Zero is no pain and 10 is the worst pain they have ever felt.
Time Frame: At time of enrollment
Population: When asking about their back pain specifically.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment for AIS | Treatment With Dynamic Myofascial Manipulation
Number analyzed (Participants) | 9 | 12
units on a scale | 2 (2.5) | 2.2 (2.1)

7. Primary Outcome: Pain Scale
Description: as for outcome 6
Time Frame: 6 months from time of enrollment
Population: When asking about their back pain specifically.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Treatment for AIS | Treatment With Dynamic Myofascial Manipulation
Number analyzed (Participants) | 8 | 10
score on a scale | 2.9 (2.5) | 1.1 (1.7)

ADVERSE EVENTS:
Time Frame: No adverse events occurred in either group from the time of enrollment to the time they completed the study which is a 6 month time frame.
Arm/Group | Standard Treatment for AIS | Treatment With Dynamic Myofascial Manipulation
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 0/9 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT05423509/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT05423509/ICF_001.pdf